CLINICAL TRIAL: NCT00492752
Title: A Randomized, Double-blinded, Placebo-controlled Study of Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11849
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Sorafenib was administered orally at a dose of 400 mg (2 x 200 mg tablets) bid (twice daily); 2 dose reductions to predefined levels of 400 mg (2 x 200 mg tablets) once daily (od) and 400 mg (2 x 200 mg tablets) every 2 days were permitted for treatment-emergent adverse events related to study treatment.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Placebo (Placebo Comparator): Placebo tablets matching in appearance were orally administered bid (twice daily).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — multikinase inhibitor; Sorafenib 400 mg (orally) twice daily
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Placebo — Matching placebo (orally) twice daily
  Arms: Placebo

SUMMARY:
The purpose of the study is

* Find out if patients receiving Sorafenib will live longer
* Find out if Sorafenib has any effect on patient reported outcomes
* Find out if Sorafenib prevents the growth or shrinks liver tumors and / or their metastases
* Determine the pharmacokinetics (PK) in patients with liver cancer

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 18 years and above, Genders eligible for study: both
* Patients who have a life expectancy of at least 12 weeks
* Patients with advanced Hepatocellular carcinoma (HCC) (unresectable, and/or metastatic) which has been histologically or cytologically documented
* Patients must have at least one tumor lesion that meets both of the following criteria

  1. Accurately measured in at least one dimension according to Response Evaluation Criteria in Solid Tumors (RECIST)
  2. Not been previously treated with local therapy
* Patients who have received local therapy, such as surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation are eligible. Previously treated lesions will not be selected as target lesions. Local therapy must be completed at least 4 weeks prior to the baseline scan
* Patients who have an Eastern Co-operative Oncology Group (ECOG) Performance Status of 0, 1, or 2

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta [Noninvasive papillary carcinoma], Tis [Carcinoma in situ: "flat tumor"]&T1 [Tumor invades subepithelial connective tissue]). Any cancer curatively treated > 3 years prior to entry is permitted
* History of cardiac disease
* Active clinically serious infections
* Known history of human immunodeficiency virus (HIV) infection
* Known central nervous system (CNS) tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2005-10; Primary Completion 2007-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- China (10):
  - Hefei, Anhui
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Nanjing, Jiangsu
  - Dalian, Liaoning
  - Hangzhou, Zhejiang
  - Beijing
  - Chongqing
  - Shanghai
  - Tianjin
- South Korea (3):
  - Seoul, Seoul Teugbyeolsi
  - Daegu
  - Seoul
- Taiwan (4):
  - Changhua
  - Tainan
  - Taipei
  - Taoyuan District

REFERENCES:
- [Result] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Result] Cheng AL, Guan Z, Chen Z, Tsao CJ, Qin S, Kim JS, Yang TS, Tak WY, Pan H, Yu S, Xu J, Fang F, Zou J, Lentini G, Voliotis D, Kang YK. Efficacy and safety of sorafenib in patients with advanced hepatocellular carcinoma according to baseline status: subset analyses of the phase III Sorafenib Asia-Pacific trial. Eur J Cancer. 2012 Jul;48(10):1452-65. doi: 10.1016/j.ejca.2011.12.006. Epub 2012 Jan 10. PMID 22240282
- [Derived] Bruix J, Cheng AL, Meinhardt G, Nakajima K, De Sanctis Y, Llovet J. Prognostic factors and predictors of sorafenib benefit in patients with hepatocellular carcinoma: Analysis of two phase III studies. J Hepatol. 2017 Nov;67(5):999-1008. doi: 10.1016/j.jhep.2017.06.026. Epub 2017 Jul 4. PMID 28687477

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with advanced hepatocellular carcinoma were enrolled from 12 Oct 2005 to 26 Jan 2007 at 23 centers in China (15 centers), Taiwan (5 centers), and Korea (3 centers).
Pre-assignment Details: 271 subjects were enrolled in a 28-day screening period; 226 subjects were randomized either to Sorafenib or placebo (2:1 ratio) (intent-to-treat [ITT] population: for efficacy analysis); 224 subjects received at least one dose of study drug (safety population: for safety analysis). Majority of screen failures did not meet the inclusion criteria.
Groups:
- A1) Sorafenib (Nexavar, BAY43-9006) - no Open Label Phase: Participants randomized to Sorafenib treatment until unblinding (August 19, 2007), Sorafenib administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid); 2 dose reductions to predefined levels of 400 mg (2 x 200 mg tablets) once daily and 400 mg (2 x 200 mg tablets) every 2 days were permitted for treatment-emergent adverse events related to study treatment.
  Note: Safety Data of participants in the arm presented here are part of the data reported in Reporting Group (RG) 1.
- A2) Sorafenib (Nexavar, BAY43-9006) - With Open Label Phase: Participants randomized to Sorafenib treatment from until unblinding (August 19, 2007) until end of trial (July 27, 2009), Sorafenib administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid); 2 dose reductions to predefined levels of 400 mg (2 x 200 mg tablets) once daily and 400 mg (2 x 200 mg tablets) every 2 days were permitted for treatment-emergent adverse events related to study treatment.
  Note: Safety Data of participants in the arm presented here are part of the data reported in Reporting Group (RG) 1.
- B1) Placebo - no Open Label Phase: Participants randomized to Sorafenib-matching Placebo until unblinding (August 19, 2007), Placebo tablets matching in appearance were orally administered twice daily (bid).
  Note: Safety Data of participants in the arm presented here are part of the data reported in Reporting Group (RG) 2.
- B2) Placebo First - Then Open Label Sorafenib Treatment Phase: Participants switched to Open-label Sorafenib treatment from Placebo after unblinding (August 19, 2007), Sorafenib administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid); 2 dose reductions to predefined levels of 400 mg (2 x 200 mg tablets) once daily and 400 mg (2 x 200 mg tablets) every 2 days were permitted for treatment-emergent adverse events related to study treatment.
  Note: Safety Data of participants in the arm presented here are the data reported in Reporting Group (RG) 3.
Period: Double Blind Treatment
Arm/Group | A1) Sorafenib (Nexavar, BAY43-9006) - no Open Label Phase | A2) Sorafenib (Nexavar, BAY43-9006) - With Open Label Phase | B1) Placebo - no Open Label Phase | B2) Placebo First - Then Open Label Sorafenib Treatment Phase
Started | 134 | 16 | 70 | 6
Received Treatment | 133 (Safety Population. 1 participant never received treatment due to an Adverse Event.) | 16 (Safety Population) | 69 (Safety Population. 1 participant never received treatment due to protocol violation.) | 6 (Safety Population)
Completed | 120 | 16 | 67 | 6
Not Completed | 14 | 0 | 3 | 0
Not completed — Death | 13 | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Period: Follow-up and/or Open Label Sorafenib
Arm/Group | A1) Sorafenib (Nexavar, BAY43-9006) - no Open Label Phase | A2) Sorafenib (Nexavar, BAY43-9006) - With Open Label Phase | B1) Placebo - no Open Label Phase | B2) Placebo First - Then Open Label Sorafenib Treatment Phase
Started | 120 | 16 | 67 | 6
Follow-up Only (no Open Label Treatment) | 120 | 0 | 67 | 0
Follow-up First, Then Open Label | 0 | 16 | 0 | 6
Completed | 34 (1 participant completed all assessments, 33 were followed up until the end of this trial) | 0 | 20 (20 participants were followed up until the end of this trial) | 0
Not Completed | 86 | 16 | 47 | 6
Not completed — Adverse Event | 0 | 2 | 0 | 2
Not completed — Death | 75 | 5 | 45 | 1
Not completed — Lost to Follow-up | 8 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Progression by clinical judgement | 0 | 1 | 0 | 2
Not completed — Radiological and clinical progression | 0 | 0 | 0 | 1
Not completed — Switch to commercial drug | 0 | 6 | 0 | 0
Not completed — Progression measurement proven | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Total
Number analyzed (Participants) | 150 | 76 | 226
Age, Continuous [Median (Full Range); unit: Years] | 51 [23 to 86] | 52 [25 to 79] | 51 [23 to 86]
Age, Customized [Number; unit: Participants]
  <65 years | 131 | 63 | 194
  >=65 years | 19 | 13 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 66 | 193
  Male | 23 | 10 | 33
Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is a scale (range 0 [fully active] to 5 [dead]) that measures how cancer affects a patient. Subjects entering this study were to have an ECOG score of 0, 1 (restricted in physically strenuous activity but ambulatory), or 2 (capable of all self care but cannot carry out work activities.
  Participants
    0 | 33 | 22 | 55
    1 | 108 | 50 | 158
    2 | 9 | 4 | 13
Tumor burden [Number; unit: Participants] — Tumor burden refers to the number of cancer cells, the size of a tumor, or the amount of cancer in the body, and is called the tumor load. Randomization was stratified by "tumor burden" assessment ie, the presence of either macroscopic vascular invasion as determined by radiological assessment and/or extra hepatic spread versus none.
  Participants
    Absent | 32 | 15 | 47
    Present | 118 | 61 | 179

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Time Frame: From randomization of the first subject until the data cut-off date approximately 23 months after start of randomization
Population: In this study the overall survival was measured for the ITT population from the date of randomization until the date of death due to any cause. For patients alive or lost to follow-up at the time of analysis, time to death was to be censored at their last date of follow-up, or at the data cut-off of 09 Aug 2007 (23 months after randomization).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 150 | 76
days | 198 [169 to 230] | 127 [114 to 166]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.014144, Log Rank; Hazard Ratio (HR) = 0.6783, 95% CI [0.4962 to 0.9272] — Hazard ratio is for Sorafenib vs placebo
Statistical Analysis 2: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.003464, Log Rank; log rank test stratified by country, tumor burden, and ECOG; Hazard Ratio (HR) = 0.6208, 95% CI [0.4498 to 0.8568] — Hazard ratio is for Sorafenib vs placebo

2. Secondary Outcome: Time to Symptomatic Progression (TTSP)
Description: Time to Symptomatic Progression (TTSP) was defined as the time from date of randomization to symptomatic progression. Subjects without symptomatic progression at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: as for outcome 1
Population: Time to Symptomatic Progression was measured for the ITT population (all randomized subjects) up to the data cut-off date of of 09 Aug 2007 (23 months after randomization)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 150 | 76
days | 105 [85 to 129] | 103 [73 to 124]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.497537, Log Rank; Hazard Ratio (HR) = 0.9032, 95% CI [0.6705 to 1.2165] — Hazard ratio is for Sorafenib vs placebo
Statistical Analysis 2: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.437926, Log Rank; log rank test stratified by country, tumor burden, and ECOG; Hazard Ratio (HR) = 0.8831, 95% CI [0.6449 to 1.2093] — Hazard ratio is for Sorafenib vs placebo

3. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) was defined as the time from date of randomization to radiologically documented disease progression. Subjects without progression at the time of analysis were censored at their last date of tumor evaluation。
Time Frame: as for outcome 1
Population: Time to progression was measured for the ITT population (all randomized subjects) up to the data cut-off date of 09 Aug 2007 (23 months after randomization).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 150 | 76
days | 84 [80 to 109] | 41.5 [41 to 47]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.000537, Log Rank; Hazard Ratio (HR) = 0.5744, 95% CI [0.4154 to 0.7942] — Hazard ratio is for Sorafenib vs placebo
Statistical Analysis 2: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.000540, Log Rank; log rank test stratified by country, tumor burden, and ECOG; Hazard Ratio (HR) = 0.5375, 95% CI [0.3763 to 0.7677] — Hazard ratio is for Sorafenib vs placebo

4. Secondary Outcome: Disease Control
Description: Disease Control (DC) was defined as the total number of subjects whose best response was not Progressive Disease (PD: an increase in the sum of tumor lesions sizes) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR: disappearance of tumor lesions) + total number of Partial Response (PR: a decrease of at least 30% in the sum of tumor lesion sizes) + total number of Stable Disease (SD: steady state of disease); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating).
Time Frame: as for outcome 1
Population: Disease control rate was measured for the ITT population (all randomized subjects)
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 150 | 76
participants
  Yes | 53 | 12
  No | 97 | 64
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006); Test type: Superiority or Other; Disease control rate = 0.3533, 95% CI [0.2771 to 0.4355]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; Disease control rate = 0.1579, 95% CI [0.0843 to 0.2596]

5. Secondary Outcome: Change in Functional Assessment of Cancer Therapy (FACT) Hepatobiliary Symptom Index-8 (FHSI-8) Score From Baseline to Cycle 1 and Cycle 3
Description: The FHSI-8 questionnaire was completed at baseline and every 3 weeks during treatment and at the end of treatment visit only for subjects who withdrew for reasons other than symptomatic progression. Patient reported outcome was measured using the FHSI-8 score changes from baseline throughout the study period. FHSI-8 assesses hepatobiliary cancer symptoms with total score ranges from 0 to 32 (0 = the best quality of life; 32 = the worst quality of life with severe symptoms)..
Time Frame: Baseline up to Cycle 1 and Cycle 3. From randomization of the first subject until the data cut-off date approximately 23 months after start of randomization
Population: FHSI-8 score changes from baseline by visit were assessed for the ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 150 | 76
scores on a scale
  cycle 1 | 26 (4.8) | 26 (4.8)
  cycle 3 | 24 (6.3) | 25 (5.3)

6. Secondary Outcome: Change in Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) Score From Baseline to Cycle 3 and End of Treatment
Description: The FACT-Hep questionnaire was also completed to assess patient reported outcome. The FACT-Hep assesses hepatobiliary cancer-related quality of life. FACT-Hep total score ranges from 0 to 180 (0=All questions answered "Not at all"; 180=All questions answered "Very much").
Time Frame: Baseline up to Cycle 3 and end of treatment. From randomization of the first subject until the data cut-off date approximately 23 months after start of randomization
Population: FACT-Hep score changes from baseline by visit were assessed for the ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 150 | 76
scores on a scale
  cycle 3 | -10 (25.5) | -3 (19.9)
  end of treatment | -25 (27.2) | -23 (31.3)

7. Secondary Outcome: Number of Participants With Different Tumor Response
Description: Tumor Response (= Best Overall Response) of a subject was defined as the best tumor response (confirmed Complete Response (CR: disappearance of tumor lesions), confirmed* Partial Response (PR: a decrease of at least 30% in the sum of tumor lesion sizes), Stable Disease (SD: steady state of disease), or Progressive Disease (PD: an increase in the sum of tumor lesions sizes)) observed during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
Time Frame: From randomization/start of treatment of the first subject until approximately 23 months after randomization when the subjects on placebo were offered the option to crossover to sorafenib treatment
Population: The tumor response was measured for the ITT population.
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 150 | 76
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 5 | 1
  Stable Disease (SD) | 81 | 21
  Progressive Disease (PD) | 46 | 41
  Not assessable | 18 | 13
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.67, Fisher Exact; based on tumor response rate (CR+PR)

8. Secondary Outcome: Duration of Response
Description: Duration of Response was defined as the time from date of first response (Complete Response (CR) or Partial Response (PR)) to the date when Progressive Disease (PD) is first documented, or to the date of death, whichever occurs first. Subjects still having CR or PR at the time of analysis were censored at their last tumor assessment.
Time Frame: as for outcome 1
Population: The duration of response was measured for the ITT population.
Measure: Median (Full Range); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 5 | 1
days | 210 [82 to 343] | 252 [252 to 252]

9. Secondary Outcome: Time to Response
Description: Time to Response (TTR) for subjects who achieved a response (Complete Response (CR) or Partial Response (PR) ) was defined as the time from date of randomization to the earliest date that the response was first documented.
Time Frame: as for outcome 1
Population: The time to response was measured for the ITT population.
Measure: Median (Full Range); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 5 | 1
days | 84 [45 to 126] | 42 [42 to 42]

10. Secondary Outcome: Area Under the Curve From Time 0 to 12 Hours Post-dose (AUC 0-12) After 21 Days of Sorafenib Treatment
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. A plot of concentration vs time after dosing is created, and the area under this curve is calculated by standard methods (eg, trapezoidal rule) to provide a measure of how much drug was in the bloodstream following dosing.
Time Frame: PK assessments made at following times: pre-dose, 1 h, 2h, 4h, 8h,and 12h after at least 21 consecutive doses during Cycle 1
Population: The stated goal in the protocol was to obtain PK data from approximately 39 patients. As this was only descriptive information, the sample size was not critical. All patients who provided PK data were included in the analysis.
Measure: Geometric Mean (Full Range); unit: mg*h/L
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 24 | 0
mg*h/L | 35.7 [7.8 to 149.2] |

11. Secondary Outcome: Normalized Area Under the Curve (AUC Norm) After 21 Days of Sorafenib Treatment
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: g*h/L
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 24 | 0
g*h/L | 6.6 [1.3 to 21.6] |

12. Secondary Outcome: Maximum Concentration (Cmax) After 21 Days of Sorafenib Treatment
Description: Cmax refers to the highest plasma concentration of drug reached after dosing. It is obtained by collecting a series of blood samples after dosing, and analyzing them for drug content by a sensitive and specific analytical method. The highest measured concentration is referred to as the Cmax.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 24 | 0
mg/L | 4.44 [1.121 to 16.7] |

13. Secondary Outcome: Normalized Maximum Concentration (Cmaxnorm) After 21 Days of Sorafenib Treatment
Description: Cmaxnorm refers to the maximum plasma concentration of Sorafenib corrected for dose and body weight (Cmaxnorm = Cmax/(mg/kg)).
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: g/mL
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 24 | 0
g/mL | 0.66 [0.18 to 2.43] |

14. Secondary Outcome: Time of Maximum Concentration (Tmax) After 21 Days of Sorafenib Treatment
Description: Tmax refers to the time after dosing when a drug attains its maximum concentration in the blood. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content. The time corresponding to the highest measurable concentration (Cmax) is referred to as Tmax.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 24 | 0
hours | 4.0 [0.5 to 12] |

ADVERSE EVENTS:
Time Frame: Reporting Group (RG) 1 + 2: Data from start of treatment until end of this trial (July 27, 2009); RG 3: Data after unblinding (August 19, 2007) until end of this trial (July 27, 2009).
Description: Acronyms in Adverse Event section: Gastrointestinal (GI), Common Terminology Criteria for Adverse Events (CTCAE), not otherwise specified (NOS), absolute neutrophil count (ANC), Central nervous system (CNS), Partial thromboplastin time (PTT), Alanine transaminase (ALT), Aspartate transaminase (AST), Gamma glutamyl transpeptidase (GGT).
Groups:
- Sorafenib, All (Double-Blind and Open Label Phase): Reporting Group 1 (RG 1): All participants randomized to Sorafenib treatment (data from start of treatment until end of trial [July 27, 2009]). Sorafenib administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid); 2 dose reductions to predefined levels of 400 mg (2 x 200 mg tablets) once daily and 400 mg (2 x 200 mg tablets) every 2 days were permitted for treatment-emergent adverse events related to study treatment.
- Placebo, All (Double-Blind and Open Label Phase): Reporting Group 2 (RG 2): All participants randomized to Sorafenib-matching Placebo (data from start of treatment until end of trial [July 27, 2009]). Treatment for Double-Blind phase (before unblinding [August 19, 2007]): Placebo tablets matching in appearance were orally administered twice daily (bid); Treatment for Open Label phase (after unblinding [August 19, 2007]): Sorafenib administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid); 2 dose reductions to predefined levels of 400 mg (2 x 200 mg tablets) once daily and 400 mg (2 x 200 mg tablets) every 2 days were permitted for treatment-emergent adverse events related to study treatment.
- Placebo, Open Label Only (Participants Switched to Sorafenib): Reporting Group 3 (RG 3): Participants switched to Open-label Sorafenib treatment from Placebo ( Data after unblinding [August 19, 2007] until end of this trial [July 27, 2009]). Sorafenib administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid); 2 dose reductions to predefined levels of 400 mg (2 x 200 mg tablets) once daily and 400 mg (2 x 200 mg tablets) every 2 days were permitted for treatment-emergent adverse events related to study treatment.
Arm/Group | Sorafenib, All (Double-Blind and Open Label Phase) | Placebo, All (Double-Blind and Open Label Phase) | Placebo, Open Label Only (Participants Switched to Sorafenib)
Serious Adverse Events (participants affected / at risk) | 76/149 | 34/75 | 3/6
Other Adverse Events (participants affected / at risk) | 144/149 | 65/75 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib, All (Double-Blind and Open Label Phase) (N=149) | Placebo, All (Double-Blind and Open Label Phase) (N=75) | Placebo, Open Label Only (Participants Switched to Sorafenib) (N=6)
Hypertension (Cardiac disorders) | 1 | 0 | 0
Cardiac General - Other (Cardiac disorders) | 0 | 1 | 0
Death Not Associated With CTCAE Term, Disease Progression NOS (General disorders) | 22 | 8 | 1
Death Not Associated With CTCAE Term, Multi - Organ Failure (General disorders) | 3 | 3 | 1
Death Not Associated With CTCAE Term, Sudden Death (General disorders) | 3 | 1 | 0
Fever (General disorders) | 5 | 3 | 0
Fatigue (General disorders) | 2 | 1 | 0
Constitutional Symptoms - Other (General disorders) | 1 | 0 | 0
Rigors / Chills (General disorders) | 1 | 0 | 0
Anorexia (Gastrointestinal disorders) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 7 | 3 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 0 | 0
Distension (Gastrointestinal disorders) | 2 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis (Functional/Symptomatic), Oral Cavity (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
GI - Other (Gastrointestinal disorders) | 2 | 1 | 0
Stricture, GI, Biliary Tree (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
CNS Hemorrhage (Vascular disorders) | 1 | 0 | 0
Hemorrhage, GI, Abdomen NOS (Vascular disorders) | 1 | 0 | 0
Hemorrhage, GI, Anus (Vascular disorders) | 0 | 1 | 0
Hemorrhage, GI, Varices (Esophageal) (Vascular disorders) | 4 | 1 | 0
Hemorrhage, GI, Stomach (Vascular disorders) | 1 | 0 | 0
Hemorrhage, GI, Liver (Vascular disorders) | 0 | 1 | 0
Hemorrhage, GI, Upper GI NOS (Vascular disorders) | 9 | 4 | 0
Hemorrhage - Other (Vascular disorders) | 1 | 0 | 0
Hemorrhage Pulmonary, Nose (Vascular disorders) | 1 | 0 | 0
Hemorrhage Pulmonary, Respiratory Tract NOS (Vascular disorders) | 0 | 1 | 0
Liver Dysfunction (Hepatobiliary disorders) | 6 | 8 | 0
Hepatobiliary - Other (Hepatobiliary disorders) | 1 | 1 | 0
Febrile Neutropenia (Infections and infestations) | 1 | 0 | 0
Infection - Other (Infections and infestations) | 2 | 1 | 0
Infection With Unknown ANC, Biliary Tree (Infections and infestations) | 0 | 1 | 0
Infection With Unknown ANC, Lung (Pneumonia) (Infections and infestations) | 4 | 1 | 0
Infection With Unknown ANC, Wound (Infections and infestations) | 1 | 0 | 0
Edema: Limb (Blood and lymphatic system disorders) | 2 | 0 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic / Lab - Other (Metabolism and nutrition disorders) | 1 | 0 | 0
CNS Ischemia (Nervous system disorders) | 2 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 3 | 0
Neuropathy: Motor (Nervous system disorders) | 1 | 0 | 0
Neurology - Other (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Syncope (Fainting) (Nervous system disorders) | 0 | 1 | 0
Pain, Back (General disorders) | 1 | 1 | 0
Pain, Chest Wall (General disorders) | 1 | 0 | 0
Pain, Tumor Pain (General disorders) | 1 | 0 | 0
Pain, Abdomen NOS (General disorders) | 7 | 3 | 0
Pain, Bone (General disorders) | 0 | 1 | 0
Pain, Other (General disorders) | 1 | 0 | 0
Pain, Pelvis (General disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Shortness of Breath) (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Renal - Other (Renal and urinary disorders) | 1 | 0 | 0
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Secondary Malignancy (Possibly Related to Cancer Treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib, All (Double-Blind and Open Label Phase) (N=149) | Placebo, All (Double-Blind and Open Label Phase) (N=75) | Placebo, Open Label Only (Participants Switched to Sorafenib) (N=6)
Allergic Reaction (Immune system disorders) | 2 | 4 | 0
Tinnitus (Ear and labyrinth disorders) | 12 | 0 | 0
Blood - Other (Blood and lymphatic system disorders) | 8 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 29 | 10 | 0
Leukocytes (Blood and lymphatic system disorders) | 18 | 4 | 0
Platelets (Blood and lymphatic system disorders) | 35 | 10 | 1
Hypertension (Cardiac disorders) | 33 | 4 | 0
PTT (Blood and lymphatic system disorders) | 12 | 4 | 0
Fatigue (General disorders) | 51 | 15 | 0
Fever (General disorders) | 38 | 8 | 0
Insomnia (General disorders) | 25 | 17 | 0
Weight Loss (General disorders) | 62 | 13 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 40 | 1 | 0
Dermatology - Other (Skin and subcutaneous tissue disorders) | 15 | 3 | 0
Hand - Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 69 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 9 | 0
Rash / Desquamation (Skin and subcutaneous tissue disorders) | 33 | 7 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Anorexia (Gastrointestinal disorders) | 46 | 13 | 0
Ascites (Gastrointestinal disorders) | 41 | 13 | 0
Constipation (Gastrointestinal disorders) | 20 | 12 | 0
Diarrhea (Gastrointestinal disorders) | 64 | 12 | 3
Distension (Gastrointestinal disorders) | 24 | 15 | 0
GI - Other (Gastrointestinal disorders) | 10 | 1 | 0
Mucositis (Clinical Exam), Oral Cavity (Gastrointestinal disorders) | 6 | 2 | 1
Nausea (Gastrointestinal disorders) | 37 | 19 | 0
Vomiting (Gastrointestinal disorders) | 25 | 13 | 0
Hemorrhage Pulmonary, Respiratory Tract NOS (Vascular disorders) | 2 | 1 | 1
Hepatobiliary - Other (Hepatobiliary disorders) | 8 | 6 | 0
Infection - Other (Infections and infestations) | 10 | 6 | 0
Edema: Limb (Blood and lymphatic system disorders) | 10 | 8 | 0
Alkaline Phosphatase (Metabolism and nutrition disorders) | 39 | 14 | 0
ALT (Metabolism and nutrition disorders) | 49 | 18 | 2
Amylase (Metabolism and nutrition disorders) | 8 | 0 | 0
AST (Metabolism and nutrition disorders) | 63 | 23 | 1
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 56 | 24 | 2
Creatinine (Metabolism and nutrition disorders) | 10 | 3 | 0
GGT (Metabolism and nutrition disorders) | 9 | 7 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 7 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 5 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 10 | 6 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 34 | 16 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 12 | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 11 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 23 | 10 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 17 | 4 | 1
Lipase (Metabolism and nutrition disorders) | 19 | 4 | 0
Metabolic / Lab - Other (Metabolism and nutrition disorders) | 33 | 9 | 0
Dizziness (Nervous system disorders) | 4 | 5 | 1
Memory Impairment (Nervous system disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 1
Optic Disc Edema (Eye disorders) | 0 | 0 | 1
Pain, Abdomen NOS (General disorders) | 54 | 16 | 0
Pain, Back (General disorders) | 23 | 9 | 0
Pain, Chest Wall (General disorders) | 12 | 2 | 0
Pain, Chest/Thorax NOS (General disorders) | 1 | 2 | 1
Pain, Dental/Teeth/Peridontal (General disorders) | 1 | 0 | 1
Pain, Head/Headache (General disorders) | 12 | 1 | 1
Pain, Joint (General disorders) | 6 | 0 | 1
Pain, Liver (General disorders) | 10 | 9 | 0
Pain, Muscle (General disorders) | 10 | 1 | 0
Pain, Other (General disorders) | 11 | 2 | 0
Pain, Stomach (General disorders) | 3 | 4 | 0
Pain, Throat/Pharynx/Larynx (General disorders) | 10 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 12 | 2
Dyspnea (Shortness of Breath) (Respiratory, thoracic and mediastinal disorders) | 17 | 12 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 11 | 7 | 0
Flu - Like Syndrome (General disorders) | 3 | 1 | 1
Pain, Bone (General disorders) | 8 | 5 | 0

LIMITATIONS AND CAVEATS:
On review of unblinded data, up to 19 Mar. 2007, the independent Data Monitoring Committee concluded the efficacy results can be considered positive, recommended subjects under placebo to cross over to Sorafenib; study continued to extension phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator must send a draft manuscript to be submitted for publication or to be presented or abstract to Bayer at least 60 days in advance of submission in order to obtain approval prior to submission of the final version for publication or presentation. In case of a difference of opinion between Bayer and the Investigator(s), the contents of the publication will be discussed in order to find a solution, which satisfies both parties.